CLINICAL TRIAL: NCT06586736
Title: The Respiratory Physiologic Efficacy of Prone Position and Its Association With Outcomes in ARDS: A Prospective Observational Cohort Study
Brief Title: Physiological Studies in the Prone Position in Patients With ARDS
Status: Recruiting | Type: Observational
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Zhou Yongfang, Principal Investigator, West China Hospital
Other Study IDs: Prone position
Record Dates: First submitted 2024-08-30; First posted 2024-09-19 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Acute Respiratory Distress Syndrome; Mechanical Ventilation; Prone Positioning
Keywords: Prone positioning; ARDS; Dead space ratio; Ventilatory ratio; Ventilation/perfusion
MeSH Terms: conditions — Respiratory Distress Syndrome; Respiratory Aspiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to observe the changes of physiological indicators such as ventilation and oxygenation in the prone position of ARDS patients, to observe the change trend of each patient's indicators, and to observe whether different trends of indicators predict different prognosis of patients.

DETAILED DESCRIPTION:
PP has been shown to effectively improve the prognosis of patients with severe ARDS, but not all patients with ARDS can benefit from PP, and the implementation of the PP has a certain clinical risks and side effects, we lack a convenient predictors to guide doctors to determine whether patients should implement the PP. Clinical usually observe the P/F improved as whether PP treatment effective reference, but there are literature points out that the rising P/F after PP can not predict the better prognosis. one of the mechanisms for ARDS patients benefit from PP is proved to be improve V/Q, the change of the V/Q may determine whether the PP treatment effectively is an important indicator. PaO2:FiO2 ratio was usually used to evaluate the effect of PP, but some studies did not support this conclusion. PP has been shown to change ventilation-perfusion ratio, dead space may be better physiological indicators, simplify dead space ratio and Ventilatory ratio can be easily accessed at bedside and is associated with mortality of patients with ARDS. The purpose of this study is to observe the predictive value of P/F, VD-etCO2/VT, and VR on the treatment effect of ARDS undergoing PP.

ELIGIBILITY:
Inclusion Criteria:

1. Intubated patients
2. Undergoing mechanical ventilation
3. Moderate to severe ARDS
4. Undergoing prone positioning
5. Age≥18 years old

Exclusion Criteria:

1. Pregnant
2. Cardiac structural shunt
3. Extracorporeal membrane oxygenation performed
4. Undergo extracorporeal CO2 removal
5. Pulmonary embolism
6. Other situation that may affect the accuracy of PetCO2 monitoring
7. Prone positioning session less than 10 hours

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We conducted a prospective cohort study in a intensive care unit in West China Hospital, Sichuan University, China. Adult patients (age≥18years) who were diagnosed with moderate to severe ARDS according to the Berlin definition, received mechanical ventilation and prone positioning were included.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
28 days without mechanical ventilation | From the date of enrollment to 28 days
  Days without mechanical ventilation support within 28 days after enrollment

SECONDARY OUTCOMES:
ICU mortality and in-hospital mortality | From the date of enrollment until the date of discharge, assessed up to 1 year
  Prognostic measures will be recorded until discharge, such as ICU mortality and in-hospital mortality
Length of lCU stay and length of hospital stay | From the date of enrollment until the date of discharge, assessed up to 1 year.
  Prognostic measures will be recorded until discharge, such as length of lICU stay and length of hospital stay in days.
Respiratory physiological parameters. | From enrollment to Day 7.
  Respiratory physiological parameters are collected at each time point (before prone positioning , every 4 hours after prone positioning, and 4 hours after turn back to supine position), such as PaO2/FiO2。
Indicators related to dead space | From enrollment to Day 7.
  Indicators related to dead space are collected at each time point (before prone positioning , every 4 hours after prone positioning, and 4 hours after turn back to supine position), such as VR and dead space ratio, which were calculated by predicted body weight, partial pressure of carbon dioxide and end-tidal carbon dioxide

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Critical care medicine of West China Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Yes
Any data collected during this study can be acquired from the correspondingauthor upon a reasonable request.
Supporting Information: CSR
Time Frame: Half a year after the publication of the research paper.
Access Criteria: Any data collected during this study can be acquired from the correspondingauthor upon a reasonable request.